CLINICAL TRIAL: NCT03801408
Title: Building Partnerships With First Responders to Explore Strategies to Improve Delivery and Access of Mental Health Services
Brief Title: Building Partnerships With First Responders to Improve Delivery and Access of Mental Health Services
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 228929
Record Dates: First submitted 2018-12-17; First posted 2019-01-11 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will conduct qualitative interviews with firefighters and EMTs/ paramedics across Arkansas. To address this aim, opt-in methods will be used to recruit a diverse group of firefighters and emergency medical technicians/paramedics from across Arkansas to participate in qualitative interviews, defined as focus groups and individual interviews. Through this work, this will generate the scientific foundation to develop a comprehensive, mental health service model that will motivate engagement in services by diverse first responders.

DETAILED DESCRIPTION:
Firefighters and emergency medical technicians (EMTs)/ paramedics respond to more than 50 million emergency calls in the U.S. every year. The daily operations and experiences that are expected and accepted as part of their job expose them to various traumatic events. The nature, frequency, and intensity of duty-related traumatic exposures place these first responders (FRs) at significant risk for mental health (MH) problems, such as post-traumatic stress disorder (PTSD) and suicide. However, due to the stigma of mental illness and the culture of self-reliance and strength that surrounds FRs, few are willing to seek help. There will be a two-stage exploratory, qualitative study that will use a statewide community-engagement approach to conceptualize a MH service model that would motivate FRs to be more engaged in services. In Stage 1, qualitative interviews with firefighters and EMTs/ paramedics will be conducted across Arkansas. In Stage 2, product development process grounded in these findings to conceptualize a MH service model feasible for implementation in real world settings. (Protocol for Stage 2 will be submitted for IRB approval at a later time.) Stage 1, Specific Aim: Identify FRs' preferences and priorities regarding MH service and delivery methods, including the feasibility, acceptability, and value of each method. To address this aim, we will use opt-in methods to recruit a diverse group of firefighters and EMTs/paramedics from across Arkansas to participate in qualitative interviews, defined as focus groups and individual interviews. After all qualitative interviews have been analyzed, a series of product development activities in Stage 2. Through this work, the scientific foundation to develop a comprehensive, MH service model that will motivate engagement in services by diverse FRs. This study's findings will guide a multi-stage, research agenda that will include development and pilot testing of the MH service model, ultimately, promoting engagement in MH services may decrease suicide rates and improve the overall MH outcomes among this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and over volunteer and career personnel active, inactive, and retired

Exclusion Criteria:

* Non- English speaking (due to the nature of focus group/interview discussions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Firefighters and EMT/paramedics in Arkansas
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Jones, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used opt-in methods, facilitated by our community partners, to recruit. The PI visited fire departments and EMS stations. The State EMS Director distributed information through the state EMS registry. Emails and promotional materials instructed first responders to contact the PI or research assistant by telephone or email for more study information. The PI was invited to present and recruit at state fire and EMS meetings. The study flyer was also placed on social media sites.
Groups:
- Arkansas First Responders: All participants were current or retired first responders in Arkansas, including certified Emergency Responders, Emergency Medical Technicians, Paramedics, and Firefighters.
Period: Overall Study
Arm/Group | Arkansas First Responders
Started | 145
Completed | 145
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arkansas First Responders
Number analyzed (Participants) | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 133
  More than one race | 1
  Unknown or Not Reported | 0
Military experience [Count of Participants; unit: Participants]
  Current military experience | 4
  Past military experience (veteran) | 19
  No military experience | 122
Department size [Count of Participants; unit: Participants]
  Small (3 or less stations) | 56
  Medium (More than 3 stations, less than 150 people) | 52
  Large (More than 150 people) | 28
  Not answered | 9
Department setting [Count of Participants; unit: Participants]
  Rural | 65
  Suburban | 10
  Urban | 25
  Mixed | 45
Previous treatment for mental health [Count of Participants; unit: Participants]
  Yes | 33
  No | 110
  Not answered | 2

OUTCOME MEASURES:

1. Primary Outcome: First Responders Who Provided Qualitative Data
Description: Number of first responders who provided perspectives and/or priorities for mental health services and/or provided suggestions for how to adapt this feedback to the population.
Time Frame: 1.5 year
Measure: Number; unit: participants
Arm/Group | Arkansas First Responders
Number analyzed (Participants) | 145
participants | 145

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Arkansas First Responders
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 0/145
Other Adverse Events (participants affected / at risk) | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03801408/Prot_SAP_000.pdf